CLINICAL TRIAL: NCT05690425
Title: A Phase I Study to Evaluate the Safety, Tolerability, Pharmacokinetics, Pharmacodynamics, and Preliminary Efficacy of BC3402 as a Single Agent in Patients With Myelodysplastic Syndrome SYNDR(MDS) and Chronic Myelomonocytic Leukemia(CMML)
Brief Title: A Phase I Study of BC3402 as a Single Agent in Patients With MDS and CMML
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Biocity Biopharmaceutics Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: BC3402-002
Record Dates: First submitted 2023-01-10; First posted 2023-01-19 (Actual); Last update posted 2023-07-24 (Actual); Status verified 2023-07

CONDITIONS: Hematologic Malignancy
Keywords: MDS and CMML
MeSH Terms: conditions — Hematologic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- BC3402 treatment group (Experimental): BC3402 as a single agent via intravenous infusion once every 3-weeks
  Interventions: Drug: BC3402 Injection

INTERVENTIONS:
Drug: BC3402 Injection — Subjects will receive BC3402 as a single agent via intravenous infusion once every 3-weeks (Q3W),the dose of BC3402 was calculated according to the dose group and body weight of the subjects.
  Other Names: not have

SUMMARY:
This is a phase I study to evaluate the safety ,Tolerability, PK, PD, and preliminary efficacy of BC3402 Monotherapy in MDS or CMML, and explore the RP2D/MTD dose.

The patients with very low,low,intermediate,or high,very high risk of MDS or CMML,who meet the criteria will receive BC3402 as a single agent via intravenous infusion Q3W , Up to 3 dose cohorts will be sequentially enrolled using an accelerated titration combined with a "3+3 design" approach.Dose limiting toxicities (DLT) will be assessed during the first cycles (i.e., total 3 weeks).

A Safety Monitoring Committee (SMC), comprised of the Sponsor's medical representatives, safety physician, and the principal investigator (PI), will be established for the determination of dose levels to be administered and dose regimen during dose escalation based on the data available from the previous dose levels. Additional dose levels may be explored based on the emerging safety, PK, and PD data during the study.

DETAILED DESCRIPTION:
This is a phase I study to evaluate the safety ,Tolerability, PK, PD, and preliminary efficacy of BC3402 Monotherapy in MDS or CMML, and explore the RP2D/MTD dose.

The patients with very low,low,intermediate,or high,very high risk of MDS or CMML,who meet the criteria will receive BC3402 as a single agent via intravenous infusion Q3W , Up to 3 dose cohorts will be sequentially enrolled using an accelerated titration combined with a "3+3 design" approach.Dose limiting toxicities (DLT) will be assessed during the first cycles (i.e., total 3 weeks). The Cohort1 will be enrolled 1 patient initially.If this subject experience any Grade 2 or higher toxicity during the first cycle, unless definitely unrelated to BC3402,2 more patients will be accrued,and the standard "3+3" dose escalation algorithm will be followed thereafter , with each cohort enrolling 3 to 6 subjects. Cohorts 2 and 3 will follow the traditional 3+3 dose escalation design. Dose limiting toxicities will be assessed during the first cycle(i.e., total21 days). If ≥ 2 subjects experience a DLT at a given dose level, the MTD would have been exceeded, further dose escalation is not pursued, and the prior dose level is expanded to six patients; if there is no more than one patient who experiences a DLT among those six patients, that dose level is considered the MTD.

A Safety Monitoring Committee (SMC), comprised of the Sponsor's medical representatives, safety physician, and the principal investigator (PI), will be established for the determination of dose levels to be administered and dose regimen during dose escalation based on the data available from the previous dose levels. Additional dose levels may be explored based on the emerging safety, PK, and PD data during the study.

ELIGIBILITY:
Inclusion Criteria:

1. The subject must be able to understand and voluntarily sign the informed consent form;
2. Subjects were 18 years old or above when they signed the informed consent form;
3. Subjects mast be willing to undergo serial bone marrow aspirate procedures on the study;
4. Morphologically confirmed diagnosis as extremely low risk, low risk, intermediate risk, high risk, extremely high risk MDS (IPSS-R classification) or CMML according to WHO (2016) diagnostic criteria, and WBC<13* 10^9/L (allowed to receive hydroxyurea or leukocyte removal before enrollment to reduce WBC count), and:

4.1 According to IPSS-R, patients diagnosis as extremely low risk, low risk or intermediate risk MDS must meet one or more of the following criteria:

1. Patients who are RBCs and/or platelets transfusion-dependent , must receive stable infusion 2U/month above for 3 months before the first dose;
2. Patients who are RBCs transfusion-dependent must Erythropoiesis stimulating agents (ESAs) failure or intolerant ;
3. Patients who are RBCs transfusion-dependent without ESA treatment mast have serum erythropoietin level >500 U/L ;
4. MDS patients with isolated del (5q) ("5q syndrome") must have disease progression or intolerance during lenalidomide treatment;
5. Platelet transfusion dependent patients must be treated with thrombopoietin receptor agonist (TPO-RA) for relapse/refractory or intolerance;
6. Persistent (>3 months) neutrophil absolute count is lower than 1.5 before screening × 10^9/L；

4.2 MDS and CMML patients rated as high-risk or extremely high-risk according to IPSS-R:

1. The monotherapy of demethylated drugs (HMA) failed (4 cycles of decitabine treatment or 6 cycles of azacytidine treatment) or was not tolerated;
2. Not suitable for intensive treatment;
3. CMML patients must fail or not tolerate at least one previous treatment (including but not limited to hydroxyurea treatment, HMA treatment, etc.);

5. Patient has an Eastern Cooperative Oncology Group(ecog) status between 0 and1;

6. Expected survival time > 3 months;

7. White blood cell count (WBC) ≤ 25 × 103/μL within 7 days prior to the first dose (hydroxycarbamide or leukapheresis is allowed to meet this criterion)

8. Platelet > 30 × 10^9/L before screening；

9. Adequate renal function:

(2) Serum creatinine ≤ 1.5 × Upper limit of normal value (ULN), and creatinine clearance ≥ 45 mL/min; If the urine protein is qualitative ≥ 2+, the 24-hour urine protein quantity shall be less than 3.5g;

10. Adequate liver function:

(3) Total serum bilirubin ≤ 1.5 × ULN (except Gilbert syndrome, this kind of subjects only meet the requirements of direct bilirubin ≤ 1.5 × ULN);

(4) Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 2.5 × ULN；

11. When screening, serum or urine pregnancy test (for female patients with fertility) was negative;

12. Patient must be a candidate for serial bone marrow aspirate and/or biopsy according to the institutions guidelines and be willing to undergo a bone marrow aspirate and/biopsy at screening, during and at the end of therapy on this study.

13. Male and female patients with fertility must agree to use medically approved contraceptive methods throughout the study period and continue to use them until 6 months after the last treatment of BC3402.

Exclusion Criteria:

1. Suitable and willing to accept hematopoietic stem cell transplantation (allogeneic or autologous);
2. Immunomodulatory drugs, including but not limited to thymosin, interleukin-2, interferon, etc., were used within 2 weeks before the first use of the test drug;
3. 3. Prior treatment with immunomodulatory agents including but not limited to thymosin, interleukin-2, and interferon within 2 weeks prior to the first dose of study drugs.
4. Patients who have used any Chinese herbal medicine or traditional Chinese medicine with anti-tumor activity within 2 weeks prior to the first dose of study drugs.
5. Patients who received live attenuated vaccine within 4 weeks prior to the first dose of study drug.
6. Prior treatment with an investigational drug within 4 weeks or 5 half-lives of the agent (whichever is longer) before the planned first dose of study drug. The washout period for biologic agents should be 28 days since the last dose.
7. Prior exposure to TIM-3 targeted therapy at any time.
8. Participants receiving chemotherapy within 14 days or 5 half lives (whichever is longer) before the first dose of study treatment;
9. Major organ surgery or significant trauma or radiotherapy within 2 weeks before entering the study;
10. Have received systemic glucocorticoid (prednisone>10mg/day or equivalent dose of the same drug) or other immunosuppressive drugs within 2 weeks before the first use of the study drug;
11. Active infections or other severe infections requiring systemic antibiotics, antiviral or antifungal drugs within 2 weeks before the first administration of the study treatment. Except for those who are treated with anti infection prevention according to local guidelines or the judgment of the researcher.
12. Known malignant tumors in progress or requiring active treatment in the past 5 years (except those diagnosed in the study). The exceptions to this exclusion criterion are as follows: basal cell carcinoma and squamous cell skin carcinoma completely resected; And completely resected carcinoma in situ of any type;
13. Active hepatitis B or C, history of HIV infection, active syphilis;
14. Patients with autoimmune diseases;
15. Known uncontrolled central nervous system (CNS) involvement;
16. Patients with history of serious cardiovascular and cerebrovascular diseases, including but not limited to, (1)Serious cardiac rhythm or conduction abnormalities, such as ventricular arrhythmia requiring clinical intervention, Ⅱ - Ⅲ degree atrioventricular block ect.

(2) During the screening period, 12 lead electrocardiogram (ECG) was measured for three times in the research center. According to the average value of the three times calculated by the QTc formula of the instrument used in the center, QTc interval> 470ms; (3) occurrence of acute coronary heart failure, acute congestive syndrome, aortic dissection, stroke or other grade 3 or above cardiovascular and cerebrovascular events within 6 months prior to the first dose of study drug (4) Patients with history of New York Heart Society (NYHA) class≥ II, or left ventricular ejection fraction (LVEF) < 50%; (5) Clinically uncontrollable hypertension

17. Mental disorders or poor compliance; 18. Patients who are being pregnant or breastfeeding. 19.Patients with other serious systemic diseases or conditions who are deemed unsuitable to participate in this clinical study at the judgement of the Investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Estimated)
Dates: Start 2023-07-06 (Actual); Primary Completion 2024-03-15 (Estimated); Study Completion 2024-06-15 (Estimated)

PRIMARY OUTCOMES:
Incidence of dose limiting toxicities(DLTs) within 28 days (first cycle) | Dose limiting toxicities (DLT) will be assessed during the first cycle (i.e., total 3 weeks).
  The DLT for this study will be evaluated in the first cycle. The DLT will include any of the following adverse events that cannot be clearly attributed to other reasons and are judged to be related to BC3402.
  1. Hematologic toxicity in the following cases:
     Hematologic toxicity ≥ grade 4 occurred in the first cycle, which could not be recovered to baseline value within 21 days after the occurrence, and bone marrow primordial cells<5%.
  2. Non hematologic toxicities:
     * Grade 2 above ALT and/or AST elevational concomitant grade 2 total bilirubin elevation(non biliary obstruction or other reasons);
     * QTcF interval > 470 ms or longer than baseline > 60 ms;
     * Grade 3 or above non-haematological toxicity;
  3. Others Any ongoing toxicity (of any grade) not caused by disease progression that results in a delay of more than 2 weeks in the next scheduled cycle;

CONTACTS AND LOCATIONS:
Overall Officials: hui zeng, prof, Principal Investigator — First Affiliated Hospital of Jinan University
Locations (1):
- The First Affiliated Hospital of Jinan University, Guangzhou, Guangdong, China